CLINICAL TRIAL: NCT02249962
Title: Option B+: ART Safety and Durability During First and Subsequent Pregnancies
Brief Title: Option B+: Study on Safety, Viral Suppression, and Survival on Second Line ART
Acronym: S4
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Ministry of Health and Population, Malawi (Other Government); University of North Carolina (Other); Lighthouse Trust (Other); Baylor College of Medicine (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: 14-1633; R01HD080485 (NIH)
Record Dates: First submitted 2014-09-11; First posted 2014-09-26 (Estimated); Last update posted 2021-03-12 (Actual); Status verified 2020-05

CONDITIONS: HIV; Infant Exposure to Efavirenz
Keywords: prospective; cohort

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum samples for:
  * HIV genotyping
  * micronutrient status
  * pharmacokinetics: efavirenz and progesterone levels for women using the contraceptive implant only
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Overall cohort: HIV+ women on Option B+ and their infants: Women (n=8000) visiting an antenatal clinic for care who will be followed prospectively for Malawi standard treatment outcomes and pregnancy outcomes as patients on Option B+
- Sub-cohort A: first HIV diagnosis: Women (n=300) who present to the antenatal care clinic and are diagnosed for the first time with HIV. These women will be started on Option B+ as anti-retroviral treatment, per Malawi Ministry of Health standard of care.
- Sub-cohort B: subsequent pregnancies failing 1st line ART: Women (n=150) who have failed first-line treatment (TDF/3TC/EFV) based on HIV RNA levels and CD4 count. These women will be switched to second-line treatment (AZT/3TC/ATZ/r) per Malawi Ministry of Health standard of care.
- Sub-cohort C: subsequent pregnancies who default from 1st line: Women (n=150) who are HIV+ and have a subsequent pregnancy who have not been adherent to first-line (Option B+: TDF/3TC/EFV). These women will be re-initiated on first-line treatment for 3 months, then evaluated to assess whether continuation on first-line treatment is sufficient, or if they need to be switched to second-line treatment (AZT/3TC/ATZ/r) per Malawi Ministry of Health standard of care.

SUMMARY:
To characterize safety, durability, antiretroviral treatment (ART) resistance, and clinical outcomes for mothers and infants exposed to the efavirenz-based Option B+ regimen for Prevention of Mother to Child Transmission (PMTCT) and HIV treatment in Malawi.

DETAILED DESCRIPTION:
Option B+ is an innovative strategy pioneered within Malawi that provides universal lifelong ART (tenofovir/lamivudine/efavirenz: TDF/3TC/EFV) for pregnant and breastfeeding women to promote maternal health and prevent HIV transmission to infants. The safety of a TDF/3TC/EFV based regimen used during pregnancy has not been systematically evaluated.

Objective 1: To characterize the long term safety, drug resistance patterns and clinical outcomes among women and their infants enrolled in the Malawi Option B+ program using TDF/3TC/EFV.

* Hypothesis 1: Over 3+ years of anticipated treatment follow-up, TDF/3TC/EFV will be associated with a toxicity rate requiring ART discontinuation of <3% and >90% virologic suppression at 36 months.
* Hypothesis 2: Women with baseline CD4 counts ≤ 350 cells/mm3 will experience greater rates of clinical events, treatment failure and ART toxicity compared to those with CD4 > 350 cells/mm3.

Objective 2: To critically evaluate women with subsequent pregnancies after initial engagement in the Option B+ Program.

Objective 2a: To determine the prevalence of treatment failure among pregnant women presenting to ANC on first-line therapy and evaluate the safety of ATZ/r based therapy among those women requiring second-line therapy.

* Hypothesis 1: HIVRNA testing at first ANC visit among women with subsequent pregnancies will demonstrate that approximately 5% of women will be failing treatment and will identify key risk factors associated with treatment failure.
* Hypothesis 2: ATZ/r based therapy during pregnancy is associated with toxicity rates requiring discontinuation in less than 5% of pregnant women.

Objective 2b: Among pregnant women defaulting from TDF/3TC/EFV, determine the treatment response to re-initiation of first-line therapy, need for second-line therapy, and characterize resistance.

- Hypothesis 1: Women re-engaging in care after program default will experience early ART treatment failure due to HIV drug resistance that developed after ART cessation during initial care.

Objective 3: To explore rates of adverse pregnancy and birth outcomes among women, presence of birth defects, and infant developmental delay among infants exposed to EFV-based ART after the first trimester (Objective 1), Efavirenz at conception (Objective 2a), and on second-line therapy with ATZ/r based ART (Objective 2a).

* Hypothesis 1: Efavirenz exposure during the first trimester is associated with a higher rate of adverse pregnancy and birth outcomes than if exposed later in pregnancy.
* Hypothesis 2: Infants exposed to EFV from first trimester will experience lower mean scores on Bayley neurodevelopment domains than those exposed later in pregnancy.

The investigators will collect data for maternal treatment outcomes, including vital status, per the national HIV program definitions: Alive, Dead, Default (>3 months since last visit), Stop, and Transfer Out. In addition to maternal treatment outcomes, the national HIV program collects data regarding the following outcomes, which the investigators will also collect: pregnancy and tuberculosis incidence after ART initiation, drug toxicity/ adverse event (Rash, Hepatitis, Lactic Acidosis, Anemia, Peripheral Neuropathy), adherence measurement (by pill count), WHO clinical stage at ART initiation, ART pharmacy refill information, and ART regimen.

ELIGIBILITY:
Inclusion Criteria:

* Female age ≥16 (includes adults and emancipated minors)
* HIV positive by 2 rapid tests approved by the Malawi Ministry of Health
* Willingness to provide informed consent

Exclusion Criteria:

* Female <16 years
* HIV negative
* Incapable of providing informed consent

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: HIV+ pregnant women and their infants recruited from three clinic sites in Lilongwe, Malawi.
Sampling Method: Non-Probability Sample
Enrollment: 12011 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with failure on Option B+ first-line treatment | Up to 36 months
  Proportion of women who fail first-line treatment as indicated by one or more of the following criteria: WHO Stage 3 or 4 events (as defined by Appendix 60 of the Adult AIDS Clinical Trials Group (AACTG)), or DAIDS grade 3 or 4 toxicity (lab serum markers), or proportion with treatment discontinuation (or death), or proportion with virologic failure (as measured by HIV RNA levels)

SECONDARY OUTCOMES:
Pharmacokinetic: progesterone level in women using contraceptive implant | months 3, 6, 12, 24
  Measure of serum progesterone and efavirenz levels among women with a contraceptive implant
Micronutrient assessment | Baseline, months 6, 12, 24, 36
Maternal CD4 count | baseline, months 12, 24, 36 post-ART initiation
  Standard of care
HIV RNA level measurement | baseline, months 3, 6, 12, 24, 36
  Standard of Care, measured to assess resistance to first-line ART
PHQ-9 evaluation | baseline, months 6, 12, 18, 24, 30, 36
  Assess maternal psychological well-being
Laboratory serum markers | baseline, months 3, 6, 9, 12, 18, 24, 30, 36
  Labs assessed include: renal function (creatinine and urinalysis), liver function, and hematology Measurements contribute to DAIDS grade 3 or 4 toxicity assessment.
Pregnancy outcome assessment | At time of pregnancy completion (birth, termination)
  Status of birth (live, stillborn, miscarriage), small for gestational age, congenital anomalies
HIV antibody testing- infant | age 1 year
Infant neuro-development assessment: Bayley score | Age 3 weeks, months 3, 6, 12, 18, 24, 30, 36
Family planning use and proportion of women with subsequent pregnancy by 36 months | Up to 36 months
  Assessing women's fertility preferences, usage of family planning methods, and pregnancy status post-ART initiation
ART Adherence: pill-count | months 3, 6, 9, 12, 18, 24, 30, 36
  Assessment of adherence to anti-retroviral medications via direct pill count at each clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Mina C Hosseinipour, MD, MPH, Principal Investigator — UNC Project- Malawi
Locations (1):
- UNC Project Malawi, Lilongwe, Malawi